CLINICAL TRIAL: NCT04350424
Title: Driving Skills Recovery Following Procedural Sedation for Gastrointestinal Endoscopy: A Prospective Cohort Study
Brief Title: Driving Skills Recovery Following Procedural Sedation for Gastrointestinal Endoscopy
Status: Terminated | Type: Observational
Why Stopped: Lack of resources and Covid-19
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, John Vargo, John J. Vargo, MD, MPH; Director Endoscopy Operations, Cleveland Clinic, The Cleveland Clinic
Other Study IDs: IRB 18-1451
Record Dates: First submitted 2019-10-24; First posted 2020-04-17 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia; Psychomotor Status
Keywords: procedural sedation; gastrointestinal endoscopy; deep sedation; moderate sedation; propofol; midazolam; fentanyl
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propofol Arm: Outpatients receiving anesthesiologist-administered propofol for elective outpatient endoscopic procedures
- Opioid / Benzodiazepine Arm: Outpatients receiving endoscopist-administered opioid / benzodiazepine for elective outpatient endoscopic procedures

SUMMARY:
This is a prospective cohort study that will analyze psychomotoric recovery using a commercially available driving simulator following sedation for endoscopic procedures in subjects undergoing elective outpatient endoscopic procedures. Patients receiving both propofol based sedation and well as those receiving a combination of fentanyl and midazolam will be studied. Baseline data will be obtained after training on the simulator. Following the procedure and after meeting standard discharge criteria, the subjects will undergo the same driving simulation to ascertain psychomotoric recovery.

DETAILED DESCRIPTION:
Procedural sedation for ambulatory endoscopy procedures is delivered millions of times per year in the United States. Current standard of care necessitates the presence of a responsible adult to take the patient from the endoscopic facility back home and to observe the patient. In addition, patients are frequently advised not to drive until the morning after the procedure. This recommendation holds true whether the procedure was performed in the morning or afternoon. Current data regarding psychomotoric recovery following procedural sedation for gastrointestinal endoscopy is quite limited. Moreover there are no data utilizing a driving simulator to gauge psychomotoric recovery in this setting.

The proposed study is a prospective, open label cohort study enrolling patients at the Cleveland Clinic's advanced endoscopy unit.

Inclusion criteria are: English speaking patients 18 years or older who currently hold a valid driver's license, are able to give informed consent and are undergoing either anesthesiologist directed propofol sedation (Group1) or a combination of an opioid and benzodiazepine targeting moderate sedation (Group 2) for elective outpatient procedures including advanced (endoscopic retrograde cholangiopancreatography, endoscopic ultrasonography, endoscopic submucosal dissection, deep enteroscopy) and non-advanced (esophagogastroduodenoscopy, colonoscopy) procedures.

Exclusion criteria include: inpatients, patients with altered mental status, legal blindness, physical limitations that would not make them candidates to be tested in the driving simulator, American Society of Anesthesiologists (ASA) ≥ 4 , urgent procedures, systolic hypotension defined as a systolic blood pressure < 90 mmHg and patients in whom English is not the primary language.

Upon enrollment the following information will be obtained: Age, gender, BMI, intended procedure, Mallampati score, medications and allergies, comorbidities (obesity, history of cardiac disease, renal insufficiency, chronic obstructive pulmonary disease, obstructive sleep apnea, diabetes mellitus, and the use of medications narcotics, antidepressants and sedatives.

Upon enrollment, the patient will undergo a 5-10 minute training session on a commercially available driving simulator. Following this, the subjects will complete a 5 minute standardized driving simulation. The subjects will then undergo their scheduled procedure.

Procedural data that will be obtained will include the type and doses of sedatives/analgesics utilized, procedure type, procedure length, use of any reversal agents or airway devices such as oropharyngeal or nasopharyngeal airways. In addition the occurrence of any intraprocedural cardiopulmonary unintended events such as hypotension, bradycardia and apnea will also be recorded.

Once the patient arrives in the recovery unit, they will be assessed every 5 minutes utilizing the observers scale for sedation and alertness (OAS). Discharge criteria would include; An OAS score of 5 (responding readily to name, with no evidence for ptosis; blood pressure and heart rate within 20% of baseline, oxygen saturation greater than 90% while breathing room air, the ability to walk without instability and the ability to drink liquids). The time from completion of the procedure to reaching the discharge criteria will be noted. At the time of reaching the discharge threshold, a repeat driving simulation will be performed utilizing the same program.

Simulator outcome variables will be analyzed by both parametric and nonparametric statistics. The variables that will be analyzed include: number of off road crashes, number of collisions with vehicles and other roadway objects, number of times over the posted speed limit, percentage of time over the posted limit, total number of times the center line was crossed, total number of times the driver went off the road, percentage of time out of lanes, overall turn signal usage, minimum distance to vehicles in drivers pedal reaction time. In addition, a summation of overall driving errors will be obtained.

An analysis comparing baseline and recovery driving simulator data within each sedation arm (anesthesiologist administered propofol or endoscopist directed opioid/benzodiazepine) will be performed. In a addition for each sedation arm, a univariate and multivariate analysis will be performed to evaluate for factors associated with delayed recovery of driving simulator performance.

ELIGIBILITY:
Inclusion Criteria:

* English speaking subjects ≥18 years
* Currently hold a valid driver's license
* Able to give informed consent
* Undergoing either anesthesiologist directed propofol sedation targeting deep sedation (Group1) or a combination of an opioid and benzodiazepine targeting moderate sedation (Group 2) for elective outpatient procedures

Exclusion Criteria:

* Inpatients
* Subjects patients with altered mental status
* Subjects with legal blindness
* Physical limitations that would not make them candidates to be tested in the driving simulator
* American Society of Anesthesiologists physical classification score ≥ 4
* Urgent procedures
* Systolic hypotension defined as a systolic blood pressure ≤ 90 mmHg
* Subjects in whom English is not a primary language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulatory subjects undergoing a variety of outpatient endoscopic procedures including advanced (ERCP, EUS, ESD, deep enteroscopy) and non-advanced (EGD, colonoscopy) procedures. Prospective, nonrandomized enrollment. Type of sedation is determined by the referring physician and not by study personnel.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Median number of summated deviations | From end of procedure until discharge, typically less than 4 hours
  Simulator Results - number of off road crashes, number of collisions with vehicles and other roadway objects, number of times over the posted speed limit, total number of times the center line was crossed, total number of times the driver went off the road, number of times turn signal not used or used inappropriately).
Center Lane Errors | From end of procedure until discharge, typically less than 4 hours
  Simulator Results - Percentage of time center lane crossed during simulated driving scenario
Median minimum distance to vehicle (feet). | From end of procedure until discharge, typically less than 4 hours
  Simulator Results - Median minimum distance to vehicle (feet) during simulated driving scenario
Mean brake pedal reaction time (seconds) | From end of procedure until discharge, typically less than 4 hours
  Simulator Results - Mean brake pedal reaction time (seconds) during simulated driving scenario

SECONDARY OUTCOMES:
Age | At baseline
  Years, (mean), Group 1 versus Group 2
Body mass index | At baseline
  kg/m2, (mean) Group 1 versus group 2
Mallampati score | At baseline
  median, Group 1 versus Group 2
Total propofol dose | From beginning to end of endoscopy, typically less than 2 hours
  mean,(mg/kg)
Total midazolam dose | From beginning to end of endoscopy, typically less than 2 hours
  mean, (mg/kg)
Total fentanyl dose | From beginning to end of endoscopy, typically less than 2 hours
  mean, (micrograms / kg)

CONTACTS AND LOCATIONS:
Overall Officials: John J Vargo, MD, MPH, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon study completion, it is anticipated that the results will be submitted for publication in a peer reviewed journal
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Bajaj JS, Heuman DM, Wade JB, Gibson DP, Saeian K, Wegelin JA, Hafeezullah M, Bell DE, Sterling RK, Stravitz RT, Fuchs M, Luketic V, Sanyal AJ. Rifaximin improves driving simulator performance in a randomized trial of patients with minimal hepatic encephalopathy. Gastroenterology. 2011 Feb;140(2):478-487.e1. doi: 10.1053/j.gastro.2010.08.061. Epub 2010 Sep 21. PMID 20849805
- [Background] Baskin-Bey ES, Stewart CA, Mitchell MM, Bida JP, Rosenthal TJ, Nyberg SL. Preliminary report of the Hepatic Encephalopathy Assessment Driving Simulator (HEADS) score. Ethn Dis. 2008 Summer;18(3):357-64. PMID 18785452